CLINICAL TRIAL: NCT02717988
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of a Single Oral Dose of SKI-O-703 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of a Single Oral Dose of SKI-O-703 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OSCO-P1201
Record Dates: First submitted 2016-03-04; First posted 2016-03-24 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; healthy volunteers; moderately to severely active
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — cevidoplenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- SKI-O-703 50 mg (Experimental): SKI-O-703 capsule (2x25 mg)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 100 mg (Experimental): SKI-O-703 capsule (4x25 mg)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 200 mg (Experimental): SKI-O-703 capsule (1x200 mg)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 400 mg (Experimental): SKI-O-703 capsule (2x200 mg)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 600 mg (Experimental): SKI-O-703 capsule (3x200 mg)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 800 mg (Experimental): SKI-O-703 capsule (4x200 mg)
  Interventions: Drug: SKI-O-703 capsule
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: SKI-O-703 capsule — SKI-O-703 25 mg capsule or 200 mg capsule without excipient
  Arms: SKI-O-703 100 mg; SKI-O-703 200 mg; SKI-O-703 400 mg; SKI-O-703 50 mg; SKI-O-703 600 mg; SKI-O-703 800 mg
Drug: Placebo capsule — Placebo 180 mg capsule filled with microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This double-blind, placebo-controlled, single ascending dose study is designed to demonstrate safety, tolerability and pharmacokinetics of SKI-O-703 in healthy volunteers. The results of this study will guide selection of dose levels for future multiple dose studies in healthy volunteers and adult patients with moderately to severely active rheumatoid arthritis.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled study in healthy adult volunteers that will be conducted to evaluate the safety, tolerability, and pharmacokinetics of ascending single doses of SKI-O-703. A total of 48 subjects are planned to participate in 6 cohorts (8 subjects each). In each cohort, 6 subjects will be randomly assigned to receive SKI-O-703 and 2 subjects will be randomly assigned to matching placebo. Dosing will be initiated in the 50 mg dose cohort and sequentially escalated to the 100 mg, 200 mg, 400 mg, 600 mg, and 800 mg cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for participation prior to completing any study procedures
* Considered by the investigator to be in good health as determined by the absence of clinically significant diseases or clinically significant abnormal values as determined by a detailed medical history review, complete physical examination, and clinical laboratory assessments. Clinical significance for any out-of-range laboratory test results will be determined by the principal investigator
* Male subjects and female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive
* Female subjects of non-childbearing potential are those who are surgically sterile at least 6 months or postmenopausal at least 2 years and have follicle-stimulating hormone serum levels consistent with postmenopausal status.
* Male subjects must agree to use a condom with spermicide or abstain from sexual intercourse for 90 days after dosing
* Male subjects must agree not to donate sperm for 90 days after dosing
* Female subjects must have negative serum pregnancy test results at Screening and Day -1
* Subject must have a body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, and weight ≥50 kg
* Subject must be able to understand the study and any risks to participation and able to communicate with the investigator

Exclusion Criteria:

* History of any clinically significant disease or disorder that may put the subject at risk if he/she participates in the study, might affect the subject's ability to participate in the study, or influence the study results
* History or presence of any gastrointestinal, hepatic or renal disease, or any other condition known to interfere with the absorption, distribution, metabolism, or excretion (ADME) of drugs
* Any surgical or medical conditions possibly affecting drug ADME (eg, bariatric procedure)
* Any medical/surgical procedure or trauma within 4 weeks of Day -1 as determined by the investigator
* Any clinically significant infection within 3 months of Day -1 as determined by the investigator
* Any of the following abnormal laboratory values upon repeat testing at Screening or check-in:

  * Hemoglobin <the lower limit of normal (LLN)
  * Platelet count <LLN
  * Absolute neutrophil count <LLN or >the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >ULN
  * Creatinine or blood urea nitrogen >ULN
  * Other clinically significant abnormal laboratory results in the opinion of the investigator
* Use of concomitant medications from 30 days or 5 half-lives prior to Day -1 (whichever is longer), including prescription medications, nutritional supplements, herbal remedies, and over-the-counter medications
* Receipt of any investigational medication within 30 days or 5 half-lives prior to Day -1, whichever is longer
* Use of tobacco or nicotine-containing products within 30 days prior to Day -1 and through the End-of-Study visit
* Use of cytochrome P450 3A isozyme (CYP3A) inducers and inhibitors (including St. John's wort) within 30 days of dosing
* Food or beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard), and charbroiled meats within 1 week prior to dosing
* History of substance abuse, drug addiction, or alcoholism
* Positive urine drug or urine alcohol test result at screening or Day -1 or unable to abstain from alcohol from 72 hours prior to study entry to the End-of-Study visit
* Unable to abstain from caffeine and xanthine-containing products from 72 hours prior to dosing through discharge from the study site
* Female subjects who are pregnant or lactating or have a positive serum pregnancy test result at Screening
* Positive test results at Screening for human immunodeficiency virus, hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, or hepatitis B core antibody and negative for HBsAg
* Recent (past 5 years) history of malignancy except successfully treated basal cell carcinoma
* High blood pressure, defined as >140 millimeters of mercury (mm Hg) systolic blood pressure or >90 mm Hg diastolic blood pressure upon repeat confirmation
* Cardiac arrhythmias or clinically significant ECG findings upon repeat confirmation by the investigator
* Corrected QT interval (QTc) >450 milliseconds or deemed clinically significant by the investigator
* Family history of long QT syndrome
* Blood loss or blood donation >450 mL within 4 weeks of study drug dosing
* History of sensitivity to drugs with chemical similarity to the study drug, its components, or excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants (Healthy Volunteers) with reported adverse events receiving single dose of SKI-O-703 as assessment of safety and tolerability. | 28 days
  Safety and tolerability of SKI-O-703 as measured by subject incidence of treatment-related Adverse Events.

SECONDARY OUTCOMES:
Area under the concentration versus time curve from time 0 to the last quantifiable concentration (AUC0-t) for estimating the pharmacokinetic parameters of SKI-O-592 (the free base of SKI-O-703) and its metabolites. | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  AUC0-t will be reported
Area under the concentration versus time curve from time 0 extrapolated to infinity (AUC0-inf) | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  AUC0-inf will be reported
Maximum observed plasma concentration (Cmax) | Days 0 (pre-dose), 1 (dosing), and post-dose at days 2, 3 and 4
  Cmax will be reported
Time to reach the maximum observed plasma concentration (Tmax) | Day 0 (pre-dose), Day1 (dosing), and post-dose at days 2, 3 and 4
  Tmax will be reported
Apparent terminal elimination half-life (T1/2) | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  T1/2 will be reported
Apparent volume of distribution (Vd/F) (SKI-O-592, free base of SKI-O-703) | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  Vd/F will be reported
Apparent oral clearance (CL/F) (SKI-O-592 only) | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  CL/F will be reported.
Terminal elimination rate constant (Kel) | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  Kel will be reported.
Mean residence time (MRT) | Day 0 (pre-dose), Day 1 (dosing), and post-dose at days 2, 3 and 4
  MRT will be reported.
Metabolite ratio (Rmet), calculated as AUC0-t (metabolite) / AUC0-t (parent) (metabolites M1, M2 and M4 only). | Day 0 (pre-dose), Day 1 (dosing) and post-dose at Days 2, 3 and 4
  Rmet will be reported.
Renal clearance (SKI-O-592, free base of SKI-O-703 only) | Day 1 (dosing), and post-dose at days 2, 3 and 4
  Renal clearance will be reported.
Amount of drug excreted in urine over the collection intervals of 0 to 4 hours (Ae0-4), 4 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 48 hours, and 48 to 72 hours post dose. | Day 1 (dosing), and post-dose at days 2, 3 and 4
  Ae will be reported

OTHER OUTCOMES:
The pharmacodynamics variable will be the change in the percentage of activated gp53/CD63+ basophils and will be evaluated from serial blood samples collected from subjects who have received SKI-O-703 or placebo. | Pre-dose, Day 1(dosing) and post-dose at Day 2
  changes in the percentage of activated gp53/CD63+ basophils will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States